CLINICAL TRIAL: NCT04244201
Title: Evaluation of Vaporous Hyperoxia Therapy (VHT) for Chronic Wounds
Brief Title: Vaporous Hyperoxia Therapy (VHT) in the Treatment of Foot Wounds
Acronym: VHT1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vaporox (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VAPOROX-VHT100-01
Record Dates: First submitted 2020-01-23; First posted 2020-01-28 (Actual); Last update posted 2020-01-30 (Actual); Status verified 2020-01

CONDITIONS: Neuropathic Foot Ulcer; Foot Ulcer
Keywords: diabetic foot; leg ulcer; skin ulcer
MeSH Terms: conditions — Foot Ulcer; Diabetic Foot; Leg Ulcer; Skin Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- VHT treatment (Experimental): Patients will be treated with VHT for 1 hour four times per week
  Interventions: Device: Vaporous Hyperoxia Therapy

INTERVENTIONS:
Device: Vaporous Hyperoxia Therapy — 1 hour of treatment, 4 times per week
  Other Names: VHT; Misty; WTS

SUMMARY:
The purpose of this study is to evaluate the effectiveness of Vaporous Hyperoxia Therapy (VHT), previously named Misty (WTS-1000) for the treatment of chronic foot ulcers.

DETAILED DESCRIPTION:
The Vaporox VHT1 study is a single arm study evaluating the efficacy of Vaporous Hyperoxia Therapy (VHT), previously named Misty (WTS-1000), as an adjunctive therapy for the treatment of chronic foot ulcers.

ELIGIBILITY:
Inclusion Criteria:

* Diabetic, arterial, and venous foot ulcers as well as decubitus ulcers
* University of Texas Health Science Center classification: Grade 0, 1, and 2

Exclusion Criteria:

* Ulcers above the medial and lateral malleoli
* Etiology of cancer/neoplastic
* Etiology of collagen vascular disease
* Etiology of gangrene
* Etiology of osteomyelitis (Grade 3)
* Etiology of thermal burns
* Etiology of radiation injury
* Pregnancy
* Acute skin conditions
* Inadequate perfusion to support treatment
* Wounds where the end cannot be probed
* Wounds covered with petroleum based dressing
* Non-compliant patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2005-06-06 (Actual); Primary Completion 2007-03-01 (Actual); Study Completion 2007-10-04 (Actual)

PRIMARY OUTCOMES:
Wound healing rate at 12 weeks | 12 weeks
  The percent of subjects that achieved wound healing at 12 weeks

SECONDARY OUTCOMES:
Time to wound healing | up to 12 weeks
  Time to achieve complete wound healing

CONTACTS AND LOCATIONS:
Overall Officials: Clifford J Wolf, DPM, Principal Investigator — Wolf Podiatry

IPD SHARING:
Plan to Share IPD: No